CLINICAL TRIAL: NCT02226666
Title: Physiologic Assessment Following Gadoxetic Acid and Gadobenate Dimeglumine Administration
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Matthew Davenport, MD, Principle Investigator, University of Michigan
Other Study IDs: HUM00075454
Record Dates: First submitted 2014-08-22; First posted 2014-08-27 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Liver Tumor
Keywords: MRI; Eovist; MultiHance
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy; gadobenic acid; gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients having MRI with Eovist: Subjects having a clinically ordered MRI with Eovist. Patients consenting for the study will be monitored before and after getting MRI contrast. For the study oxygen saturation (amount of oxygen level in the blood) and breathing will be monitored during the can. Breathing will be measured with a non-invasive respiratory monitoring device attached to the MR scanner. Each patient will answer survey questions after the scan about their experiences concerning MRI contrast.
  Interventions: Drug: MRI with Eovist
- Patients having MRI with Multihance: Subjects having a clinically ordered MRI with Multihance. Patients consenting for the study will be monitored before and after getting MRI contrast. For the study oxygen saturation (amount of oxygen level in the blood) and breathing will be monitored during the scan. Breathing will be measured with a non-invasive respiratory monitoring device attached to the MR scanner. Each patient will answer survey questions after the scan about their experiences concerning MRI contrast.
  Interventions: Drug: MRI with Multihance

INTERVENTIONS:
Drug: MRI with Multihance — Patients will have Multihance used as an IV contrast agent for their scan.
  Other Names: gadobenate dimeglumine
  Groups: Patients having MRI with Multihance
Drug: MRI with Eovist — Patients will have Eovist used as an IV contrast agent for their scan.
  Other Names: Gadoxetate disodium
  Groups: Patients having MRI with Eovist

SUMMARY:
The purpose of this study is to prospectively compare the physiologic response of patients who receive either intravenous gadoxetic acid (Eovist) or intravenous gadobenate dimeglumine (MultiHance).

DETAILED DESCRIPTION:
Contrast-enhanced hepatic MRI is an accepted method for detecting and characterizing liver lesions. Liver lesion characterization is fundamental for patient management, because lesions that meet specific imaging criteria for hepatocellular carcinoma (HCC) are assumed to be HCC without tissue confirmation. There are a variety of gadolinium-based contrast agents that are used for this purpose. Two of the more commonly utilized are gadoxetic acid (an hepatobiliary contrast agent that permits 20 minute hepatobiliary phase imaging) and gadobenate dimeglumine (a weak hepatobiliary contrast agent that functions generally as an extracellular contrast agent). A recent study by our group has shown that patients who receive intravenous gadoxetic acid are much more likely to experience transient dyspnea after contrast injection that causes them to breathe rapidly through the arterial phase of imaging, degrading image quality. In that study, subjective complaints of dyspnea and respiratory motion artifact on imaging were scored. The investigators did not assess patient physiologic response. The goal of the proposed work is to build on our prior data and to determine whether there are non-invasively measurable physiologic parameters that can support our original study. Specifically, the investigators want to determine whether there are predictable changes in SpO2, pulse, respiratory periodicity, and respiratory regularity that correlate with arterial phase image degradation and patients complains of dyspnea. Both contrast agents to be assessed in this study are FDA approved with at least 4 years of post-marketing experience documenting safety and efficacy. The investigators will not be changing or altering our clinical approach in any way as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older
* Patients scheduled for MRI examination at the University of Michigan hospital
* Patients receiving either MultiHance or Eovist contrast agents during their clinical MRI examination

Exclusion Criteria:

* Patients under 18 years of age
* Patients who will not receive MultiHance or Eovist as part of their clinical MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One-hundred patients receiving gadoxetic acid for hepatobiliary indications and 100 patients receiving gadobenate dimeglumine for hepatobiliary indications will be studied prospectively. All patients will be scheduled to undergo MRI for clinical purposes by their primary care physicians. The patients will not be randomized.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Survey | Baseline
  Subjects fill out a short 5-question survey about their MRI experience directly following clinical MRI scan.

SECONDARY OUTCOMES:
Oxygen Levels | Baseline
  We will monitor a subjects' oxygen levels by placing a small monitor on one of their fingers before and after the MRI; lasting approximately one minute each.
Respiratory Rate | Baseline
  We will monitor a subjects' respiratory rate (how many times they breathe in a minute) during the clinical MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davenport, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No